CLINICAL TRIAL: NCT02099448
Title: Correlation of Non-invasive Assessment, Using C.A 2.0 Device, Versus Invasive Assessment of Left Ventricular End Diastolic Pressure (LVEDP)
Brief Title: Correlation of Non-invasive Assessment, Using C.A 2.0 Device, Versus Invasive Assessment of LVEDP
Status: Completed | Type: Observational
Sponsor: CorAlert Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: COR-01
Record Dates: First submitted 2014-03-26; First posted 2014-03-28 (Estimated); Last update posted 2016-02-09 (Estimated); Status verified 2016-02

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Elective Cardiac Catheterization

SUMMARY:
The purpose of the study is to determine the accuracy of non-invasive assessment of LVEDP using the investigational device C.A 2.0.

ELIGIBILITY:
Inclusion Criteria:

1. Male subject between the ages of 18 - 80 years or postmenopausal female up to 80 years of age
2. Patient undergoing elective cardiac catheterization during which LVED and aortic pressures are recorded
3. Willing and able to sign informed consent prior to study initiation

Exclusion Criteria:

1. Subject has a baseline heart rate of < 60 or >100 beats/min
2. Subject has moderate to severe valvular disease
3. Subject suffers from atrial fibrillation or other tachyarrhythmias
4. Subject suffers from hemodynamic instability
5. Subject is candidate for primary PCI

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects undergoing elective cardiac catheterization, during which LVED and aortic pressures are recorded
Sampling Method: Non-Probability Sample
Enrollment: 41 (Actual)
Dates: Start 2014-04; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Establish the accuracy of the non-invasive device, C.A 2.0, to estimate LVEDP comparing it to the invasive hemodynamic measurement via left heart catheterization | During elective cardiac catheterization

CONTACTS AND LOCATIONS:
Locations (1):
- Kaplan Medical Center, Rehovot, Israel